CLINICAL TRIAL: NCT06350162
Title: A Randomized Controlled, Multicenter Phase II Study to Evaluate the Efficacy and Safety of Combination Therapy With Serplulimab and RT in Patients With ES-SCLC Who Have Not Progressed After Treat With Serplulimab Combined Chemotherapy
Brief Title: Testing the Addition of Radiation Therapy to the Immune Therapy Treatment for ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Fan Yun, MD, Head of Chest Oncology Department, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASTRUM-LC12
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Extensive Stage Lung Small Cell Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serplulimab+Radiation Therapy (Experimental): Patients receive Serplulimab IV over 30 minutes +/- 10 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo radiation therapy QD on days 1-5 during weeks 1-3 only. Patients undergo PET/CT scan, CT, and MRI throughout the trial. Patients also undergo blood and tissue collection throughout the trial.
  Interventions: Drug: Serplulimab; Radiation: Chest Radiation
- Serplulimab (Active Comparator): Patients receive Serplulimab IV over 30 minutes +/- 10 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo PET/CT scan, CT, and MRI throughout the trial. Patients also undergo blood and tissue collection throughout the trial.
  Interventions: Drug: Serplulimab

INTERVENTIONS:
Drug: Serplulimab — 4.5mg/kg,IV over 30 minutes +/- 10 minutes on day 1. Cycles repeat every 21 days.
  Other Names: HLX10
Radiation: Chest Radiation — 30Gy-45Gy/QD/3Gy
  Arms: Serplulimab+Radiation Therapy

SUMMARY:
This phase II trial compares the effect of adding radiation therapy to the usual maintenance therapy with Serplulimab versus Serplulimab alone in patients who have already received Serplulimab plus chemotherapy for the treatment of extensive stage small cell lung cancer .

DETAILED DESCRIPTION:
This phase II trial compares the effect of adding radiation therapy to the usual maintenance therapy with Serplulimab versus Serplulimab alone in patients who have already received Serplulimab plus chemotherapy for the treatment of extensive stage small cell lung cancer . Immunotherapy with monoclonal antibodies, such as Serplulimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving radiation therapy in addition to Serplulimab may extend the time without extensive small cell lung cancer growing or spreading compared to Serplulimab alone.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical studies; fully understand, be informed about the study and have signed the informed consent form (ICF).
2. Male or female aged ≥ 18 and ≤ 75 years, at the time of signing the ICF.
3. Willingness to follow and ability to complete all trial procedures.
4. Histologically or cytologically diagnosed with ES-SCLC (according to the Veterans Administration Lung Study Group staging system).
5. No prior systemic therapy for ES-SCLC；at the end of the combination chemotherapy with serplulimab, the efficacy evaluation is CR, PR, or SD.
6. At least one measurable lesion as assessed according to RECIST 1.1 , lesions that have received radiation therapy in the past are only considered measurable if they show clear progression.
7. An ECOG PS score of 0 or 1.
8. An expected survival ≥ 3 months.
9. Normal major organ functions
10. For participants receiving therapeutic anticoagulation: stable anticoagulant regimen
11. Negative human immunodeficiency virus (HIV) test at screening
12. Negative hepatitis B surface antigen (HBsAg) test at screening
13. Positive hepatitis B surface antibody (HBsAb) test at screening, and positive hepatitis B virus core antibody (HBcAb), no HBV-DNA test is required; or negative HBsAb at screening accompanied by either of the following: Negative total hepatitis B core antibody (HBcAb), or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test. The HBV DNA test will be performed only for participants who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test.
14. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for participants who have a positive HCV antibody test.
15. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception.
16. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm.

Exclusion Criteria:

1. Complete response or tumor progression occurred during the combination of serplulimab and chemotherapy treatment.
2. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.Patients with CNS lesions treated and Asymptomatic are eligible to participate in this study if they meet all of the following criteria: Measurable lesions exist outside of CNS that meet the definition of RECISTv1.1; The patient has no history of Intracranial hemorrhage or intracerebral hemorrhage; The patient did not receive stereotactic radiotherapy within 7 days before the start of the study treatment, whole brain radiotherapy within 14 days before the start of the study treatment, or Neurosurgery resection within 28 days before the start of the study treatment; Patients do not need to continue to receive Corticosteroid treatment for CNS diseases. Allowing stable doses of anticonvulsant drugs for treatment; Transfer is limited to the cerebellum or supratentorial area (i.e. not transferred to the midbrain, pons, medulla oblongata, or spinal cord); There is no evidence to suggest progress between the completion of CNS local treatment and the initiation of study treatment; New Asymptomatic patients with central nervous system metastasis found during screening are eligible to participate in this study after receiving radiotherapy and/or surgery
3. History of leptomeningeal disease.
4. The total number of liver metastases was ≥3 or a single liver metastases was greater than 3cm
5. Uncontrolled tumor-related pain
6. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
7. Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN).
8. Known active or suspected autoimmune diseases. Subjects in a stable state with no need for systemic immunosuppressant therapy are allowed to enroll.
9. Have a history of Idiopathic pulmonary fibrosis, organized pneumonia (such as Bronchiolitis obliterans), drug-induced pneumonia or idiopathic pneumonia, or chest computed tomography (CT) at screening shows evidence of active pneumonia.
10. Active or latent pulmonary tuberculosis.
11. Serious cardiovascular disease (such as heart disease, myocardial infarction or cerebrovascular accident of New York Heart Association Grade II or above), unstable arrhythmia or unstable angina pectoris occurred within 3 months before the start of the study treatment.
12. Major surgical procedures other than diagnosis have been performed within 4 weeks prior to the start of the study treatment, or significant surgical procedures are expected to be required during the study period.
13. Malignant tumors other than small cell lung cancer (SCLC) occurred within 5 years before the start of the study treatment, but the cancer under study and malignant tumors with negligible risk of metastasis or death (such as the 5-year overall survival rate>90%) were excluded, such as fully treated cervical Carcinoma in situ, non Melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ or stage I Uterine cancer.
14. Severe infection occurred within 4 weeks before the start of study treatment, including but not limited to hospitalization due to infection, Bloodstream infections, severe pneumonia or any active infection that may affect the safety of patients.
15. Previously received allogeneic stem cell or solid organ transplantation.
16. Any other diseases, metabolic disorders, physical examination abnormalities, or clinical laboratory abnormalities that may affect the interpretation of results or treatment complications that may pose a high risk to patients, may result in contraindications to the use of research drugs.
17. Received attenuated live vaccines within 4 weeks prior to the start of research treatment, or expected to receive such vaccines during the treatment period of sulumab or within 5 months after the last administration of serplulimab.
18. Currently undergoing anti HBV treatment.
19. Received any other investigational drug treatment within 28 days prior to the start of the study treatment.
20. Previous treatment with CD137 agonists or immune checkpoint blockade therapy, including anti CTLA-4, anti PD-1, and anti PD-L1 therapeutic antibodies.
21. Received systemic immunostimulatory therapy (including but not limited to interferon and interleukin-2 [IL-2]) within 4 weeks prior to the start of study treatment or within 5 drug elimination half-lives (whichever is longer).
22. Systemic immunosuppressive drugs (including but not limited to Corticosteroid, Cyclophosphamide, Azathioprine, methotrexate, Thalidomide and anti TNF - α preparations) were used within 2 weeks before the start of the study treatment, or systemic immunosuppressive drugs were expected to be used during the study treatment, with the following exceptions: 1)Patients receiving short-term, low-dose systemic immunosuppressive drugs or patients receiving one-time pulse therapy of systemic immunosuppressive drugs (for example, receiving Corticosteroid for 48 hours to treat contrast allergy) may be qualified to participate in this study after being confirmed by the medical supervisor; 2) Patients who receive Mineralocorticoid (such as fluhydrocortisone), inhaled or low-dose Corticosteroid to treat Chronic obstructive pulmonary disease (COPD) or asthma, or low-dose Corticosteroid to treat orthostatic Hypotension or adrenal insufficiency are eligible to participate in this study.
23. Has a history of severe allergies to chimeric or humanized antibodies or fusion proteins.
24. Known hypersensitivity to serplulimab.
25. Known hypersensitivity to carboplatin or etoposide.
26. Pregnant or lactating women, or women who plan to become pregnant during the study treatment or at least 5 months after the last administration of Slulimab or 6 months after the last administration of cisplatin/carboplatin or Etoposide.
27. Researchers determine that patients cannot benefit from TRT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year Progression-free survival rate | up to 1year
  PFS rate after 1 year after randomization

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months after last patient randomized
  defined as time from randomization to the date of first observed disease progression (investigator assessment according to RECIST 1.1) or death from any cause
Overall survival (OS) | up to 22 months after last patient randomized
  defined as the time from initiation of study treatment to death from any cause
Duration of response (DOR) | up to approximately 24 months
  defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Disease control rate (DCR) | up to approximately 24 months
  defined as the proportion of participants who have a best overall response of CR or PR or stable disease (SD), as determined by the investigator according to RECIST v1.1.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From baseline up to approximately 24 months
  An adverse event was defined as any untoward medical occurrence in a participant

CONTACTS AND LOCATIONS:
Overall Officials: Yun Fan, PHD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No